CLINICAL TRIAL: NCT06833957
Title: PReparing for OptimalPhase III/IV maTErnal Group B StreptococCal Vaccine Trials in Africa (PROTECT)
Brief Title: Preparing for Maternal GBS Vaccine Trials in Africa
Acronym: PROTECT
Status: Recruiting | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Fundação Manhiça (Other); Universiteit Antwerpen (Other); LINQ Management GMBH (Unknown); Aga Khan University (Other); University of Liverpool (Other); Kamuzu University of Health Sciences (Other); MU-JHU CARE (Other); St George's, University of London (Other); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 101145724
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-01

CONDITIONS: Group B Streptococcus; Invasive Bacterial Diseases (IBD); Maternal Immunization
Keywords: Child health; Clinical research; Clinical trials; Infectious diseases; Group B Streptococcus; vaccines; maternal immunisation; maternal health
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- WP2: Pregnancy Episode Registries: This work package (WP2) will develop systems to determine background pregnancy and infancy outcomes, as defined by Global Alignment of Immunization Safety Assessment in Pregnancy (GAIA), in preparation for maternal vaccine clinical trials and post-implementation studies. WP2 will assess the utility of existing medical records data to accurately determine pregnancy events following immunisation and, using patient data related to atleast 4000 pregnancies in each country, to establish an easy to use pregnancy episodes registry (PER) that can be used for future Phase III/IV trials. The PER will be developed using freely available code developed under EDCTP2 so that it can be used in other African settings in the future.
  The WP2 group consists of pregnant women and their infants up to hospital discharge at the chosen health facilities in Uganda, Malawi, Mozambique, and Kenya.
- WP3: GBS disease sentinel site surveillance: WP3 will conduct a prospective observational GBS surveillance study among infants less than 90 days old who are admitted with laboratory confirmed GBS at sentinel sites in Kenya, Uganda, Malawi and Mozambique. The WP3 study team will develop and strengthen IBD surveillance, with a focus on GBS in each site. All of the proposed sites have access to microbiological capacity that will be leveraged to monitor microbiologically confirmed neonatal sepsis burden. In doing so, WP3 will improve the nations' ability to participate in late phase clinical trials and post-licensure effectiveness studies in preparation for phase III/IV GBS maternal vaccine clinical trials and vaccine decision making.
  The WP3 group consists of all infants less than 90 days old admitted with GBS infection detected in blood or cerebrospinal fluid (CSF) by culture, or GBS detected in CSF by quantitative polymerase chain reaction, at the health facilities in the four countries during a period of at least 12 months.
- WP4: Vaccine confidence: Many low- and middle-income countries face significant challenges regarding vaccine implementation including vaccine confidence and participation in vaccine clinical trials, especially for vaccines targeting pregnant women. Through a mixed-methods study, WP4 will assess the knowledge, attitudes and practices of pregnant women, health care providers, community members and other relevant stakeholders towards maternal vaccines, and assess the understanding and willingness to participate in maternal vaccine trials in Kenya, Malawi, Mozambique and Uganda. WP4 will also co-create a communication/education toolkit to enhance understanding of the importance of maternal vaccines and participation in maternal vaccine trials.
  The WP4 group therefore consists of pregnant women and health care workers at the identified health facilities at the time of fieldwork. It will also consist of stakeholders such as Ministries of Health, community leaders, religious, political, or cultural leaders.

SUMMARY:
Infections are one of the key causes of newborn deaths. Among them, Group B Streptococcus (GBS) is the leading cause of sepsis and bacterial meningitis in the first 90 days of life.

Fortunately, GBS vaccines for pregnant women, a powerful tool for fighting infections, are currently in development. Once vaccine trials are completed, these vaccines can stop preventable newborn deaths.

The PReparing for Optimal Phase III/IV maTErnal Group B StreptococCal vaccine Trials in Africa (PROTECT) project, funded by the European & Developing Countries Clinical Trials Partnership (EDCTP) and European Commission, is supporting medical sites in Kenya, Malawi, Mozambique, and Uganda to establish uniform pregnancy and infant health data collection processes. It is also establishing surveillance of GBS in newborns to determine incidence rates and measure the burden of disease. With better reporting systems, medical sites can participate in vaccine trials and monitor vaccine safety. At the same time, the consortium is working to understand the drivers of vaccine hesitancy and to develop culturally appropriate communication tools to facilitate engagement with vaccines.

The end goal is to set up a network of sites that can monitor vaccine safety for current and future vaccines.

DETAILED DESCRIPTION:
Two vaccines designed for pregnant women, to protect their unborn infant, are entering late phase development and will prevent infections from GBS and respiratory syncytial virus, respectively. For these vaccines to be approved, the vaccine must work effectively without causing any unwanted responses. To implement these vaccines in countries with low resources, healthcare systems must be strengthened by improving vaccine safety monitoring and surveillance of infection, and advancing vaccine delivery, vaccine confidence, and patient participation.

The PROTECT study, funded by the EU Commission EDCTP, is three-fold:

1. Establishment of pregnancy exposure registries:

   The rapid rollout of electronic health records (EHR) in some East African countries offers an opportunity to use routine data to strengthen reporting of rates of adverse pregnancy, neonatal and infant outcomes, and any adverse events following immunisation; this will be imperative in informing and preparing for future large scale vaccination rollout campaigns. The approach will develop pregnancy registries embedded within national reporting systems to establish this data, including baseline rates of pregnancy and infancy outcomes for Tetanus and COVID19 vaccines currently in use. These reporting systems will allow monitoring of potential safety signals once new vaccines are introduced.
2. Developing sentinel site GBS microbiological surveillance:

   The investigators will conduct a prospective observational GBS surveillance study among infants less than 90 days old who are admitted with laboratory confirmed GBS. The investigators will develop and strengthen invasive bacterial disease (IBD) surveillance, with a focus on GBS in Kenya, Malawi, Mozambique and Uganda. Each of the proposed lead sites has access to microbiological capacity that will be leveraged to monitor microbiologically confirmed neonatal sepsis burden. In doing so, the investigators will improve the nations' ability to participate in late phase clinical trials and post-licensure effectiveness studies.
3. Vaccine Confidence:

The aim of this study is evaluating the knowledge and practices of pregnant women and other key stakeholders around vaccination and factors influencing vaccine confidence during pregnancy. The investigators will also create tools and communication strategies to improve willingness of pregnant women to participate in vaccine trials and consequently increase confidence in vaccines and vaccine trials during pregnancy in Mozambique, Uganda, Malawi and Kenya.

The investigators will work closely with the World Health Organization (WHO), African Medicines Agency and Country Stakeholders. This programme of work culminates in a network of maternal vaccine trial sites that can rapidly evaluate vaccines in pregnancy from late-stage trials through to introduction on a national level.

ELIGIBILITY:
Inclusion Criteria:

* WP2 Pregnancy Exposure Registries inclusion criteria:

All women and their infants attending for antenatal and/or delivery and postpartum services at the study sites in Uganda, Malawi, Mozambique, and Kenya.

WP3 GBS Surveillance inclusion criteria:

* Infants aged less than 90 days old with laboratory-confirmed GBS infection admitted at participating health facilities in Uganda, Malawi, Mozambique, and Kenya.
* Infants whose parents or guardians provided written informed consent for their participation.
* Residents in the catchment area of participating health facilities.

WP4 Vaccine Confidence inclusion criteria:

* In Uganda, Kenya and Mozambique, pregnant women at any gestation period aged 18 years and above (reproductive age).
* In Malawi, pregnant women aged 16 years are eligible to be included in the study because they are considered emancipated minors.
* Pregnant women who consent to the study and give written consent.
* Stakeholders who include pregnant women, health workers, women leaders, community leaders, national stakeholders, cultural and religious leaders who are willing to take part and can give written informed consent.

Exclusion Criteria:

WP4 Vaccine Confidence exclusion criteria:

* Pregnant women who are visiting/non-resident in the research area.
* Those who may be unwell and unable to consent to take part in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: WP2 Pregnancy Exposure Registries study population:
  Pregnant women and their infants up to hospital discharge at the chosen health facilities in Uganda, Malawi, Mozambique, and Kenya.
  WP3 GBS surveillance study population:
  All infants less than 90 days old admitted with GBS infection detected in blood or CSF by culture, or GBS detected in CSF by qPCR, at referral health facilities in the four countries during a period of at least 12 months.
  WP4 study population:
  All pregnant women attending the identified health facilities at the time of fieldwork and the health care workers who provide services to these women. It will also consist of stakeholders including, but not limited to, health workers from each country's Ministry of Health, head of facilities, community leaders (community gatekeepers and influencers), older women who give support in the community, male leaders, religious, political, administrative or cultural leaders.
Sampling Method: Non-Probability Sample
Enrollment: 18100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Pregnancy exposure registries outcome 1.1 | 01.03.2026 - 28.02.2027
  To establish pregnancy episode registries at sentinel site locations, at least 1 - 3 sites per country.
Pregnancy exposure registries outcome 1.2 | 01.03.2026 - 28.02.2027
  To generate longitudinal cohort data on pregnancies, deliveries and infant outcomes for maternal vaccine safety assessment, specifically rates of obstetric and neonatal outcomes as defined by the GAIA project.
Pregnancy exposure registries outcomes 1.3 | 01.03.2026 - 28.02.2027
  To generate comparable essential data across Kenya, Malawi, Mozambique and Uganda on adverse pregnancy, neonatal and infant outcomes using consensus definitions for maternal vaccine safety assessment.
Sentinel site GBS disease surveillance outcome 2.1 | 01.01.2025 - 01.09.2025
  To develop and strengthen capacities for GBS disease surveillance in infants less than 90 days old at sentinel sites in four African countries, using microbiological and molecular detection methods.
Sentinel site GBS disease surveillance outcome 2.2 | 01.03.2026 - 28.02.2027
  To determine the incidence rates of early and late onset iGBS disease among infants less than 90 days old admitted across established sentinel sites.
Vaccine confidence outcome 3.1 | 01.03.2025 - 28.02.2027
  To enhance understanding of the importance of vaccination in pregnancy.
Vaccine confidence outcome 3.2 | 01.03.2025 - 28.02.2027
  To understand willingness to participate in maternal vaccine trials in the four countries.
Vaccine confidence outcome 3.3 | 01.11.2025 - 20.08.2026
  To co-develop an educational/communication toolkit with key stakeholders to enhance understanding of the importance of maternal vaccines in pregnancy in the four countries.

SECONDARY OUTCOMES:
Sentinel site GBS disease surveillance outcome 2.3 | 01.09.2025 - 28.02.2027
  To assess the antimicrobial resistance patterns of GBS isolates among infants less than 90 days old.
Sentinel site GBS disease surveillance outcome 2.4 | 01.09.2025 - 28.02.2027
  To determine the genomic profile of iGBS strains.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Nakabembe, Study Director — MU-JHU CARE
Locations (9):
- Kenya (2):
  - Mariakani Sub-County Hospital, Mariakani, Coast
  - Rabai Sub County Hospital, Rabai, Kilifi County
- Malawi (3):
  - Queen Elizabeth Central Hospital, Blantyre, Blantyre District
  - Lirangwe Health Centre, Blantyre, Blantyre District
  - Ndirande Health Centre, Blantyre, Blantyre
- Mozambique (3):
  - Hospital Geral De Mavalane, Maputo, Cidade de Maputo
  - Jose Macamo General hospital, Maputo, Cidade de Maputo
  - Manhiça District Hospital, Manhiça, Manhiça
- Kawempe National Referral Hospital, Kampala, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
As soon as possible following study completion, CSG and ISGlobal will deposit the de-identified datasets in access-controlled data repositories. CSG will use Figshare (https://knowledge.figshare.com/about), and ISGlobal will use the Consortium for Catalan Universities (CSUC) and CERCA public repository (https://dataverse.csuc.cat/dataverse/ISGlobal). DOIs will be created for the datasets. Interested scientists will thus be able to see what the metadata are and can contact CSG and ISG to gain access for research purposes.
  The genome sequences will be held on Genebank, in addition to the sequencing data and associated metadata being made publicly available in research repositories such as the European Nucleotide Archive.
Time Frame: Anticipated start date: 01/05/2027 No end date.
Access Criteria: Scientists interested in the PROTECT data will be able access the IPD to view the metadata in the public research repositories and Genebank.
  The data collected in this project will be quantitative data generated from clinical assessments and medical records (entered onto digital clinical report forms -CRF- via the REDCap secure database); microbiological data, molecular data and whole genome sequences.
  Scientists interested in the PROTECT data will be able to view the metadata in the public research repositories and Genebank. Following an access request they will be able to view the associated data.

REFERENCES:
- [Background] Bramugy J, Mucasse H, Massora S, Vitorino P, Aerts C, Mandomando I, Paul P, Chandna J, Seedat F, Lawn JE, Bardaji A, Bassat Q. Short- and Long-term Outcomes of Group B Streptococcus Invasive Disease in Mozambican Children: Results of a Matched Cohort and Retrospective Observational Study and Implications for Future Vaccine Introduction. Clin Infect Dis. 2022 Jan 20;74(Suppl_1):S14-S23. doi: 10.1093/cid/ciab793. PMID 34725690
- [Background] Paul P, Chandna J, Procter SR, Dangor Z, Leahy S, Santhanam S, John HB, Bassat Q, Bramugy J, Bardaji A, Abubakar A, Nasambu C, Libster R, Yanotti CS, Seedat F, Horvath-Puho E, Hossain AKMT, Sadeq-Ur Rahman Q, Jit M, Newton CR, Milner K, Goncalves BP, Lawn JE; GBS long term outcomes LMIC collaborative group. Neurodevelopmental and growth outcomes after invasive Group B Streptococcus in early infancy: A multi-country matched cohort study in South Africa, Mozambique, India, Kenya, and Argentina. EClinicalMedicine. 2022 Apr 28;47:101358. doi: 10.1016/j.eclinm.2022.101358. eCollection 2022 May. PMID 35747160
- [Background] Aerts C, Leahy S, Mucasse H, Lala S, Bramugy J, Tann CJ, Madhi SA, Bardaji A, Bassat Q, Dangor Z, Lawn JE, Jit M, Procter SR. Quantifying the Acute Care Costs of Neonatal Bacterial Sepsis and Meningitis in Mozambique and South Africa. Clin Infect Dis. 2022 Jan 20;74(Suppl_1):S64-S69. doi: 10.1093/cid/ciab815. PMID 34725702
- [Background] Goncalves BP, Procter SR, Paul P, Chandna J, Lewin A, Seedat F, Koukounari A, Dangor Z, Leahy S, Santhanam S, John HB, Bramugy J, Bardaji A, Abubakar A, Nasambu C, Libster R, Sanchez Yanotti C, Horvath-Puho E, Sorensen HT, van de Beek D, Bijlsma MW, Gardner WM, Kassebaum N, Trotter C, Bassat Q, Madhi SA, Lambach P, Jit M, Lawn JE; GBS Danish and Dutch collaborative group for long term outcomes; GBS Low and Middle Income Countries collaborative group for long term outcomes; GBS Scientific Advisory Group, epidemiological sub-group; CHAMPS team. Group B streptococcus infection during pregnancy and infancy: estimates of regional and global burden. Lancet Glob Health. 2022 Jun;10(6):e807-e819. doi: 10.1016/S2214-109X(22)00093-6. Epub 2022 Apr 28. PMID 35490693
- [Background] Absalon J, Simon R, Radley D, Giardina PC, Koury K, Jansen KU, Anderson AS. Advances towards licensure of a maternal vaccine for the prevention of invasive group B streptococcus disease in infants: a discussion of different approaches. Hum Vaccin Immunother. 2022 Dec 31;18(1):2037350. doi: 10.1080/21645515.2022.2037350. Epub 2022 Mar 3. PMID 35240933
- [Background] Moon S, Bermudez J, 't Hoen E. Innovation and access to medicines for neglected populations: could a treaty address a broken pharmaceutical R&D system? PLoS Med. 2012;9(5):e1001218. doi: 10.1371/journal.pmed.1001218. Epub 2012 May 15. PMID 22615544
- [Background] Rottingen JA, Chamas C, Goyal LC, Harb H, Lagrada L, Mayosi BM. Securing the public good of health research and development for developing countries. Bull World Health Organ. 2012 May 1;90(5):398-400. doi: 10.2471/BLT.12.105460. No abstract available. PMID 22589577
- [Background] Philip RK, Shapiro M, Paterson P, Glismann S, Van Damme P. Is It Time for Vaccination to "Go Viral"? Pediatr Infect Dis J. 2016 Dec;35(12):1343-1349. doi: 10.1097/INF.0000000000001321. PMID 27626913
- [Background] Mehta U, Clerk C, Allen E, Yore M, Sevene E, Singlovic J, Petzold M, Mangiaterra V, Elefant E, Sullivan FM, Holmes LB, Gomes M. Protocol for a drugs exposure pregnancy registry for implementation in resource-limited settings. BMC Pregnancy Childbirth. 2012 Sep 3;12:89. doi: 10.1186/1471-2393-12-89. PMID 22943425
- [Background] Boytchev H. Maternal RSV vaccine: Further analysis is urged on preterm births. BMJ. 2023 May 10;381:1021. doi: 10.1136/bmj.p1021. No abstract available. PMID 37164373
- [Background] Chaithongwongwatthana S, Yamasmit W, Limpongsanurak S, Lumbiganon P, Tolosa JE. Pneumococcal vaccination during pregnancy for preventing infant infection. Cochrane Database Syst Rev. 2015 Jan 23;1(1):CD004903. doi: 10.1002/14651858.CD004903.pub4. PMID 25613573
- [Background] Salam RA, Das JK, Dojo Soeandy C, Lassi ZS, Bhutta ZA. Impact of Haemophilus influenzae type B (Hib) and viral influenza vaccinations in pregnancy for improving maternal, neonatal and infant health outcomes. Cochrane Database Syst Rev. 2015 Jun 9;2015(6):CD009982. doi: 10.1002/14651858.CD009982.pub2. PMID 26059051
- [Background] Giles ML, Krishnaswamy S, Macartney K, Cheng A. The safety of inactivated influenza vaccines in pregnancy for birth outcomes: a systematic review. Hum Vaccin Immunother. 2019;15(3):687-699. doi: 10.1080/21645515.2018.1540807. Epub 2018 Nov 15. PMID 30380986
- [Background] Ginsburg AS, Klugman KP. Vaccination to reduce antimicrobial resistance. Lancet Glob Health. 2017 Dec;5(12):e1176-e1177. doi: 10.1016/S2214-109X(17)30364-9. Epub 2017 Nov 8. No abstract available. PMID 29128252
- [Background] Yusuf N, Raza AA, Chang-Blanc D, Ahmed B, Hailegebriel T, Luce RR, Tanifum P, Masresha B, Faton M, Omer MD, Farrukh S, Aung KD, Scobie HM, Tohme RA. Progress and barriers towards maternal and neonatal tetanus elimination in the remaining 12 countries: a systematic review. Lancet Glob Health. 2021 Nov;9(11):e1610-e1617. doi: 10.1016/S2214-109X(21)00338-7. PMID 34678200
- [Background] Marchant A, Sadarangani M, Garand M, Dauby N, Verhasselt V, Pereira L, Bjornson G, Jones CE, Halperin SA, Edwards KM, Heath P, Openshaw PJ, Scheifele DW, Kollmann TR. Maternal immunisation: collaborating with mother nature. Lancet Infect Dis. 2017 Jul;17(7):e197-e208. doi: 10.1016/S1473-3099(17)30229-3. Epub 2017 Apr 19. PMID 28433705
- [Background] Lawn JE, Bianchi-Jassir F, Russell NJ, Kohli-Lynch M, Tann CJ, Hall J, Madrid L, Baker CJ, Bartlett L, Cutland C, Gravett MG, Heath PT, Ip M, Le Doare K, Madhi SA, Rubens CE, Saha SK, Schrag S, Sobanjo-Ter Meulen A, Vekemans J, Seale AC. Group B Streptococcal Disease Worldwide for Pregnant Women, Stillbirths, and Children: Why, What, and How to Undertake Estimates? Clin Infect Dis. 2017 Nov 6;65(suppl_2):S89-S99. doi: 10.1093/cid/cix653. PMID 29117323
- See also: PROTECT study website — https://www.protect-network.org/